CLINICAL TRIAL: NCT04516603
Title: Randomized Placebo-controlled Phase II Cross-over Study on the Influence of Fampridine on Working Memory in Healthy Subjects
Brief Title: Influence of Fampridine on Working Memory in Healthy Subjects
Acronym: Fampyr_2020
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Changement of study design. Restart spring 2021. See new registration number: NCT04652557 (FamH)
Sponsor: Prof. Dominique de Quervain, MD (Other)
Collaborators: Clinical Trial Unit, University Hospital Basel, Switzerland (Other); University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Prof. Dominique de Quervain, MD, Director Division of Cognitive Neuroscience, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2020-01626
Record Dates: First submitted 2020-08-11; First posted 2020-08-18 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Working Memory
MeSH Terms: interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fampridine SR (Experimental): Single oral administration of a tablet fampridine (10 mg) formulated for oral administration taken once in the morning without food. Tablets must be administered whole.
  The single intake is followed by a washout period of at least 7 days equalling over 40 half-lives of the active substance fampridine (t½ = 3.61 h) between experimental and control intervention.
  Interventions: Drug: Fampridine SR
- Placebo (Placebo Comparator): Identically looking placebo tablets consisting of the identical additives formulated for oral administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fampridine SR — Fampridine is an inhibitor of voltage-gated potassium (Kv) channels and is approved in Switzerland for treatment of gait problems in patients with Multiple Sclerosis (MS).
  Arms: Fampridine SR
Drug: Placebo — no active component
  Arms: Placebo

SUMMARY:
Proof-of-concept study on the effects of 10 mg fampridine (oral administration) on working memory in healthy participants.

The hypotheses is that fampridine improves working memory performance.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* generally healthy
* normotensive (BP between 90/60 mmHg and 140/90 mmHg)
* BMI between 19 and 29,9 kg/m2
* aged between 18 and 30 years
* fluent German-speaking
* Informed consent as documented by signature

Exclusion Criteria:

* contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to 4-aminopyridine
* use of potassium channel blockers within the last 3 months
* concomitant treatment with OCT 2 inhibitors (e.g. cimetidine, propranolol)
* acute or chronic psychiatric disorder (e.g. major depression, psychoses, somatoform disorder, suicidal tendency)
* acute cerebrovascular condition
* history of seizures
* risk of lowered seizure threshold (due to e.g. sleep deprivation, withdrawal of alcohol after alcohol abuse)
* renal impairment
* history of malignant cancers
* walking problems (e.g. due to dizziness)
* other clinically significant concomitant disease states (e.g. hepatic dysfunction, cardiovascular disease, diabetes, asthma)
* clinically significant laboratory or ECG abnormality that could be a safety issue in the study
* known or suspected non-compliance
* drug or alcohol abuse
* inability to follow the procedures of the study, e.g. due to language or psychological problems of the participant
* participation in another study with an investigational drug within the 30 days preceding and during the present study
* prior participation (less than two years ago) in a study investigating working memory (notably the n-back task)
* enrolment of the investigator, his/her family members, employees and other dependent persons
* smoking (>3 cigarettes per day)
* intake of psychoactive drugs (e.g. benzodiazepines, antidepressants, neuroleptics)
* pregnancy or breast feeding

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2040-01-01 (Estimated); Primary Completion 2041-12-31 (Estimated); Study Completion 2041-12-31 (Estimated)

PRIMARY OUTCOMES:
Medium-load working memory performance | test day 1 and 2, each 4 hours after intake of study medication to assess differences between the Verum and Placebo condition
  Accuracy as assessed by a letter n-back task (Papassotiropoulos, Henke et al. 2011) with the levels 0-back and 2-back.
  This test includes a 2-back task assessing working memory and a 0-back task ('x-target' task) measuring concentration. The 2-back task requires participants to respond to a letter repeat with one intervening letter (for example, S-m-s-g…). The 'x-target' task requires participants to respond to the occurrence of the letter 'x' in a sequence of letters (for example, N-l-X-g…). Accuracy (i.e. correct 2-back responses minus correct 0-back responses) will be calculated.

SECONDARY OUTCOMES:
Reaction time | test day 1 and 2 each 4 hours after intake of study medication to assess differences between the Verum and Placebo condition
  Reaction time for correct 2-back responses minus correct 0-back responses.
N-back with a 3-back condition | test day 1 and 2 each 4 hours after intake of study medication to assess differences between the Verum and Placebo condition
  N-back with a 3-back condition, which is more demanding than the 2-back condition. Accuracy (3-back minus 0-back) will be calculated.
Symbol Digit Modalities Test, SDMT | test day 1 and 2 each 4 hours after intake of study medication to assess differences between the Verum and Placebo condition
  Symbol Digit Modalities Test, SDMT (Smith 2013, 13th edition), a processing speed test. The test consists of the presentation of a series of 9 symbols, each of them is paired with a single digit, labeled 1-9, in a key at the top of a sheet. The remainder of the page has a pseudorandomized sequence of the symbols and the participant must respond with the digit associated with each of these as quickly as possible. The score is the number of correct answers in 90 seconds. The administration of SDMT will be preceded by a learning sequence at both timepoints. A parallel version will be used for the second test day.
Bochumer Matrizentest (BOMAT - advanced -short) | test day 1 and 2 each 4 hours after intake of study medication to assess differences between the Verum and Placebo condition
  Bochumer Matrizentest (BOMAT - advanced -short; Hossiep/Turck/Hasella, 2001, 1st edition), matrix reasoning. The BOMAT will be administered to measure fluid intelligence (Gf) consisting of 29 items. A time-limited version will be used according to Jaeggi (Jaeggi 2010). The total score is calculated by summing the correct solutions, ranging between 0 to 29. A parallel version will be used for the second test day.
Digit Span Task | test day 1 and 2 each 4 hours after intake of study medication to assess differences between the Verum and Placebo condition
  Digit span task, a subtest of the "Wechsler Intelligenztest für Erwachsene" (WIE;von Aster 2006). Total scores for digit span forward and backward will be calculated as described in the manual of the WIE. A parallel version will be used for the second test day.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique de Quervain, Prof, Study Chair — University of Basel, Transfaculty Research Platform; Andreas Papassotiropoulos, Prof, Study Chair — University of Basel, Transfacutly Research Platform
Locations (1):
- University of Basel, Transfaculty Research Platform, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All IPD (de-identified) that underlie results in a publication will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be available after publication, study protocol (including statistical analysis plan) will be made available before start of the study.
Access Criteria: All IPD (de-identified) that underlie results in a publication will be shared upon reasonable request for scientific purposes. A reasonable request consists of a short description of the scientific purpose. Requests will be reviewed by the team of the principle investigator.